CLINICAL TRIAL: NCT04934943
Title: "Mini Fluid Challenge Assessment: a Comparison Among Three Hemodynamic Tools"
Acronym: MINI3
Status: Not yet recruiting | Type: Observational
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: MINI3
Record Dates: First submitted 2021-06-11; First posted 2021-06-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Sepsis; Shock, Septic; Critically Ill
Keywords: Fluid challenge; Functional hemodynamic test
MeSH Terms: conditions — Sepsis; Shock, Septic; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intervention _mini_FC: The fluid challenge consists of 4 ml*Kg of Crystalloids' solution infused over 10 minutes, administered via either a central or a peripheral line.
  1. The patient is already connected to the PICCO monitoring for clinical purpose of hemodynamic monitoring (before study enrollment)
  2. The MOSTCARE system is connected to the MONITOR of the patient (and not to the patient itself) by means of a cable inserted into the connections system.
  3. The echocardiography will be performed by a senior intensivist/cardiologist. The stroke volume is calculated by measuring VTI and diameter at the same point. This is best performed by measuring the diameter of the LVOT in the parasternal long axis (PLAX) view
  Interventions: Diagnostic Test: mini_FC

INTERVENTIONS:
Diagnostic Test: mini_FC — 100 ml of Crystalloids infused over 1 minute - data recording and new baseline - FC 4 ml/kg in 10 minutes - data recording

SUMMARY:
The mini fluid challenge (mini_FC) is a functional hemodynamic test which has been used in different clinical contexts to assess fluid responsiveness.

This test is performed by rapidly injecting a small aliquot of fluid (100 ml over 1 minute), which is followed by the infusion of the residual aliquot of fluid.

Since the threshold of the mini_FC identified by the literature is rather small (5% of stroke volume (SV) increase after the 100 ml bolus to discriminate between responder and non-responder), it is crucial that the hemodynamic tool assessing this change could be reliable. Moreover, the SV changes with inspiratory/expiratory movements and the increase after the mini_FC should also consider the physiological fluctuations of the SV.

In the literature this test has been performed by means of tolls with different least significant change of the SV. The least significant change (LSC) represents the smallest difference between successive measurements of SV that can be considered to be a real change and not attributable to chance.

The purpose of this study is to assess the agreement among MOSTCARE system (4.5& of SV LSC described in the literature) and the echocardiography (about 10% of SV LSC described in the literature) with the PICCO system (about 1% of SV LSC described in the literature - considered the gold standard) in discriminating fluid responsiveness after a mini_FC

DETAILED DESCRIPTION:
Targeted fluid therapy has received increasing attention in the management of patients showing acute circulatory failure in both intensive care unit (ICU) and operating room (OR), aiming at preventing both inadequate tissue blood flow and fluid overload. In fact, unnecessary fluid administration can increase morbidity and mortality and length of hospital stay of critically ill and surgical patients.

Since the only physiological reason to give a fluid challenge (FC) is to increase the stroke volume (SV) and this effect is obtained only in about 50% of ICU and OR patients, a vast literature investigated the possibility of predict this effect before FC administration, but the issue remains extremely challenging. Bedside clinical signs and pressure and static volumetric static variables, do not predict fluid responsiveness. Moreover, several physiological factors affect the reliability of the ventilator-induced dynamic changes in pulse pressure and stroke volume [pulse pressure variation (PPV) and stroke volume (SV) variation (SVV), respectively], and their echographic surrogates, in a significant number of ICU and OR patients.

To overcome these limitations, the functional hemodynamic assessment (i.e. the assessment of the dynamic interactions of hemodynamic variables in response to a defined perturbation), of fluid responsiveness has gained in popularity. A functional hemodynamic test (FHT) consist in a manoeuvre determining a sudden change in cardiac function and/or heart lung interaction, affecting the hemodynamics of fluid responders and non-responders to a different extent.

The FHT called passive leg raising (PLR) has been successfully used for assessing the fluid responsiveness in ICU patients since 2009 and its reliability has been confirmed by three large meta-analyses. However, the PLR is not usually practicable in the OR.

A lot of different FHTs have been proposed, as alternative to the PLR, in ICU and, more recently, OR. These tests could be basically subdivided in two groups. A subgroup of FHTs is based on sudden and brief variations of the mechanical ventilation to induce a change in right ventricle preload and/or after load and, as consequence, of left ventricle. Among these tests, the rapid administration of a small aliquot of the predefined FC (the so-called mini FC) has gained in popularity in the last years.

On of the drawbacks of this test is that the optimal threshold identified in the literature to stratify responders and non-responders (5% of SV variation) is quite small, and potentially affected by the reliability of the hemodynamic tool used. The aim of this paper is to compare the reliability of a hemodynamic invasive tool (the (PiCCO2 TM, Pulsion Medical Systems, Munich, Germany - considered the gold standard) with a mini-invasive tool (MostCareTM system (Vytech Health, Padua, Italy) and a non-invasive (echocardiography) in predicting the response to the mini-FC in critically ill patients.

ELIGIBILITY:
Inclusion criteria

1) Acute circulatory failure defined as:

* SAP ≤ 90 mmHg (or a decrease > 50 mm Hg in hypertensive patients)
* or a mean arterial pressure (MAP) ≤ 70 mmHg
* or the use of vasopressors to maintain SAP >90 mmHg,
* associated with skin mottling; tachycardia ≥100 beats/min; urinary flow ≤0.5 mL/kg for at least 2 hours; blood lactate level ≥4 mmol/L.

Exclusion criteria:

* known severe myocardial or valvular dysfunction
* cardiac arrhythmias
* severe acute respiratory distress syndrome
* on-going haemodialysis or continuous hemofiltration
* moribund patients
* persistent low quality of the arterial signal affecting hemodynamic monitoring measurements
* poor echographic windows.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults critically ill patients with acute circulatory failure, who require volume expansion decided by the clinician in charge.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Agreement of allocation | immediately after the procedure
  Number of responders and non-responders identified by the MOSTCARE and the Echocardiography with respect to the PICCO system (considered as gold standard)

SECONDARY OUTCOMES:
Least significant change of the stroke volume - PICCO | 5 minutes before FC administration
  off-line analysis of the recorded stroke volume change before the test
Least significant change of the stroke volume - MOSTCARE | 5 minutes before FC administration
  off-line analysis of the recorded stroke volume change before the test
Least significant change of the stroke volume - Echocardiography | 5 minutes before FC administration
  off-line analysis of the recorded stroke volume change before the test
ROC curve - PICCO | 1 minute after mini fluid challenge infusion
  ROC curve analysis of stroke volume changes after mini fluid challenge infusion
ROC curve - MOSTCARE | 1 minute after mini fluid challenge infusion
  ROC curve analysis of stroke volume changes after mini fluid challenge infusion
ROC curve - Echocardiograhy | 1 minute after mini fluid challenge infusion
  ROC curve analysis of stroke volume changes after mini fluid challenge infusion
Agreement stroke volume estimation - MOSTCARE versus PICCO | immediately after the procedure
  Agreements between stroke volume data are determined using the Bland-Altman method, with the bias calculated as the mean difference between methods and reflecting the measurement error between the two tests.
Agreement stroke volume estimation - Echocardiography versus PICCO | immediately after the procedure
  Agreements between stroke volume data are determined using the Bland-Altman method, with the bias calculated as the mean difference between methods and reflecting the measurement error between the two tests.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Humanitas Research Hospital, Rozzano, MILANO
  - Antonio Messina, Novara, Novara

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Messina A, Lionetti G, Foti L, Bellotti E, Marcomini N, Cammarota G, Bennett V, Saderi L, Sotgiu G, Della Corte F, Protti A, Monge Garcia MI, Romagnoli S, Cecconi M. Mini fluid chAllenge aNd End-expiratory occlusion test to assess flUid responsiVEness in the opeRating room (MANEUVER study): A multicentre cohort study. Eur J Anaesthesiol. 2021 Apr 1;38(4):422-431. doi: 10.1097/EJA.0000000000001406. PMID 33399372
- [Background] de Courson H, Ferrer L, Cane G, Verchere E, Sesay M, Nouette-Gaulain K, Biais M. Evaluation of least significant changes of pulse contour analysis-derived parameters. Ann Intensive Care. 2019 Oct 11;9(1):116. doi: 10.1186/s13613-019-0590-z. PMID 31602550
- [Background] Georges D, de Courson H, Lanchon R, Sesay M, Nouette-Gaulain K, Biais M. End-expiratory occlusion maneuver to predict fluid responsiveness in the intensive care unit: an echocardiographic study. Crit Care. 2018 Feb 8;22(1):32. doi: 10.1186/s13054-017-1938-0. PMID 29415773
- [Background] Messina A, Dell'Anna A, Baggiani M, Torrini F, Maresca GM, Bennett V, Saderi L, Sotgiu G, Antonelli M, Cecconi M. Functional hemodynamic tests: a systematic review and a metanalysis on the reliability of the end-expiratory occlusion test and of the mini-fluid challenge in predicting fluid responsiveness. Crit Care. 2019 Jul 29;23(1):264. doi: 10.1186/s13054-019-2545-z. PMID 31358025
- [Background] Shi R, Monnet X, Teboul JL. Parameters of fluid responsiveness. Curr Opin Crit Care. 2020 Jun;26(3):319-326. doi: 10.1097/MCC.0000000000000723. PMID 32332283
- [Background] Vistisen ST, Scheeren TWL. Challenge of the Mini-fluid Challenge: Filling Twice without Creating a Self-fulfilling Prophecy Design. Anesthesiology. 2018 May;128(5):1043-1044. doi: 10.1097/ALN.0000000000002141. No abstract available. PMID 29664782
- [Background] Biais M, de Courson H, Lanchon R, Pereira B, Bardonneau G, Griton M, Sesay M, Nouette-Gaulain K. Mini-fluid Challenge of 100 ml of Crystalloid Predicts Fluid Responsiveness in the Operating Room. Anesthesiology. 2017 Sep;127(3):450-456. doi: 10.1097/ALN.0000000000001753. PMID 28640019